CLINICAL TRIAL: NCT07125235
Title: Reactive Driven Support for Treatment, Adherence, Resilience, and Thriving (reSTART) mHealth Randomized Controlled Hybrid Type I Effectiveness Implementation Trial
Brief Title: Reactive Driven Support for Treatment, Adherence, Resilience, and Thriving (reSTART) Clinical Trial
Acronym: reSTART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Florida International University (Other); San Diego State University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-44467; UH3DA058304 (NIH)
Record Dates: First submitted 2025-08-01; First posted 2025-08-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Behavioral Intervention; Viral Suppression of HIV Infection; ART Adherence
Keywords: HIV; Stimulant Use; mHealth
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Controlled Hybrid Type I Effectiveness Implementation Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- reSTART Intervention (Experimental): The reSTART intervention will be administered to this group and includes: (1) adherence self-monitoring tools delivered during a single baseline motivational interviewing session; (2) the urine tenofovir point-of-care self-test with adherence feedback and visualizations with motivational messages; (3) a positive affect intervention delivered via a mobile health application which supports stimulant-using men in reducing stimulant use.
  Interventions: Behavioral: reSTART Objective Adherence Self-Monitoring and Postive Affect mHealth Intervention; Device: urine tenofovir point-of-care self-test
- Standard of Care (No Intervention): The control group will receive standard of care and will not receive the reSTART intervention.

INTERVENTIONS:
Behavioral: reSTART Objective Adherence Self-Monitoring and Postive Affect mHealth Intervention — The reSTART intervention integrates a mobile health application, a urine tenofovir point-of-care self-test, and adherence feedback with motivational messages to increase HIV medication intake, reduce stimulant use, and improve HIV virologic suppression.
  Other Names: Reactive Driven Support for Treatment, Adherence, Resilience, and Thriving (reSTART)
  Arms: reSTART Intervention
Device: urine tenofovir point-of-care self-test — urine tenofovir point-of-care self-test
  Arms: reSTART Intervention

SUMMARY:
Men who are living with HIV and use stimulants face many challenges and barriers that may interfere with remembering to take their HIV medication. Forgetting to take HIV medication puts men living with HIV at a greater risk of becoming virally unsuppressed. Researchers are doing this study to test if a remote intervention can help participants improve remembering to take their HIV medications and reduce the HIV viral load among men living with HIV who use stimulants.

DETAILED DESCRIPTION:
A resurgent stimulant epidemic among men living with HIV could compromise the U.S. Ending the HIV Epidemic goals by interfering with HIV care engagement, adherence, and virologic suppression among men living with HIV. Prominent multi-level factors interfere with HIV virologic suppression for men living with HIV, particularly among those who use stimulants. This study is a nested randomized clinical trial to test a multi-component intervention to improve virologic suppression, adherence, and stimulant use among men living with HIV who use stimulants. The intervention, known as reSTART, will combine an evidence-based positive affect mobile health (mHealth) intervention, a home-based urine point-of-care test for adherence self-monitoring, and motivational interviewing and messages. The goal of the reSTART intervention is to improve or maintain adherence to HIV medications and reduce stimulant use. By this high-impact study's end, the investigators will have identified the impact of a multi-component reSTART mHealth intervention using novel point-of-care adherence self-monitoring on HIV virologic suppression and stimulant use.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed antiretroviral therapy (ART) with a tenofovir-based regimen.
* Documented virologic non-suppression, urine tenofovir testing without tenofovir detected, or self-reported adherence <100%.
* Reports stimulant use.
* Has a mailing address within the U.S.
* Currently has a smartphone with photo capabilities.

Exclusion Criteria:

* Have any health condition that may interfere with participation or the ability to provide informed consent, including any debilitating or life-threatening conditions.
* Not prescribed ART.
* Unwilling to perform urine self-testing or to attend a local Quest site for viral load monitoring.
* Unable to provide a hair sample of ~50-100 strands of hair that are non-gray, not bleached, and at least 1cm in length

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Viral suppression measured by HIV-1 RNA, Quantitative, Real-Time PCR | Baseline to 6-months post-intervention
  The primary endpoint will be change in viral suppression comparing baseline to post-intervention viral load results measured by HIV-1 RNA, Quantitative, Real-Time PCR. Viral suppression is defined as viral load results that yield less than 50 copies/mL.

SECONDARY OUTCOMES:
Stimulant Use measured quantitatively by stimulant levels in hair | Baseline to 6-months post-intervention
  Stimulant levels will be compared pre- and post-intervention and measured quantitatively using liquid chromatography-mass spectrometry laboratory techniques.
Long-term Viral Suppression measured by HIV-1 RNA, Quantitative, Real-Time PCR. | Baseline to 12-months post-intervention
  As a secondary endpoint, long-term viral suppression will be measured at 12-months and compared to baseline viral load results from HIV-1 RNA, Quantitative, Real-Time PCR. Viral suppression is defined as viral load results that yield less than 50 copies/mL.
Adherence to Tenofovir-based antiretroviral therapy | Baseline to 6-months post-intervention
  Urine tenofovir levels measured by the urine tenofovir point-of-care self-test lateral flow assay at baseline and 6-months post-intervention will be compared to assess the presence or absence of tenofovir and changes in adherence to HIV medications.

OTHER OUTCOMES:
Acceptability of the Intervention using the Theoretical Framework of Acceptability Questionnaire | Enrollment to 6-months post-intervention
  The acceptability of the intervention will be measured using the Theoretical Framework of Acceptability Questionnaire. Questions will be framed using Likert scales where a score of 1 corresponds to completely unacceptable and a score of 5 corresponds to completely acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Spinelli, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No